CLINICAL TRIAL: NCT01885897
Title: IL-15 Super Agonist ALT-803 to Treat Relapse Of Hematologic Malignancy After Allogeneic Stem Cell Transplantation
Brief Title: IL-15 Super Agonist ALT-803 to Treat Relapse Of Hematologic Malignancy After Allogeneic SCT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012LS023; HM2013-12 (Other: University of Minnesota Blood and Marrow Transplant Program)
Record Dates: First submitted 2013-06-11; First posted 2013-06-25 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-07

CONDITIONS: Acute Myelogenous Leukemia (AML); Acute Lymphoblastic Leukemia (ALL); Myelodysplastic Syndromes (MDS); Lymphoma; Myeloma; Chronic Lymphocytic Leukemia (CLL); Chronic Myelogenous Leukemia (CML)
Keywords: Acute myelogenous leukemia (AML); Acute lymphoblastic leukemia (ALL); Myelodysplastic syndromes (MDS); Lymphoma; Myeloma; Chronic Lymphocytic Leukemia (CLL); Chronic myelogenous leukemia (CML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma; Neoplasms, Plasma Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study treatment (Experimental): Weekly dose of ALT-803 at assigned dose, ranging from 1mcg/kg to 30 mcg/kg (based on phase 1 dose escalation schedule,) IV once a week for 4 weeks.
  Interventions: Biological: ALT-803

INTERVENTIONS:
Biological: ALT-803 — Given weekly IV at assigned dose level, ranging from 1mcg/kg to 30mcg/kg.

SUMMARY:
This is a multi-center, phase I/II clinical trial for patients who have relapsed more than 60 day after allogeneic transplant for a hematologic malignancy. The study consists of two phases. The dose finding phase is a modified version of a phase I trial and the extended phase is a modified version of a phase II trial.

The primary objective of the dose finding phase is to determine the maximum tolerated, minimum efficacious dose (MTD/MED) of a interleukin-15 (IL-15) super agonist complex (ALT-803) when given once weekly for 4 weeks in the outpatient setting. The study will follow a standard 3+3 design of dose escalation for toxicity with an added feature of stopping early if efficacy is confirmed. There are six dose levels of ALT-803 for to determine the MTD/MED: 1, 3, 6, 10, 20, and 30 mcg/kg.

Once the MTD/MED for ALT-803 is determined, this cohort will be used in the extended phase. The primary goal of this extended phase is to study the potential efficacy of ALT-803 in this patient population. Efficacy will be measured using rates of remission induction. An optimal Simon's two-stage design will be used in this phase. Stage 1 will enroll 14 patients (including the 6 patients treated at the MTD/MED during the dose finding phase). If 3 or more of these 14 patients respond to ALT-803, the trial will move to stage 2 and enroll an additional 23 patients. If 2 or fewer respond, the study will terminate enrollment early.

ELIGIBILITY:
Inclusion Criteria:

* Relapse after previous allogeneic stem cell transplant for one of the following hematologic malignancies (acute myelogenous leukemia, acute lymphoblastic leukemia,myelodysplastic syndromes, lymphoma, myeloma, Chronic lymphocytic Leukemia, chronic myelogenous leukemia):

  * For non-CML, relapse will be defined based on disease specific morphologic criteria from a bone marrow biopsy and aspirate or recurrence of disease specific cytogenetics. For disease specific definition of relapse, see appendix III. Relapse can be determined morphologically. Equivocal results for relapse should result in a repeated test after an appropriate time interval (suggested 1 month) to determine eligibility.
  * For CML, relapse will be defined as any cytogenetic evidence of a Philadelphia chromosome or persistence of BCR/ABL rearrangements by molecular testing on at least two measurements over a 6 month interval. If cytogenetics are normal and there is PCR evidence of a BCR/ABL fusion, patients will be eligible if they have evidence of a quantitative increase in CML measured either by quantitative PCR or by fluorescent in situ hybridization (FISH).

For Chronic Phase CML patients only:

* must have failed (no response in 3 months or incomplete response at 6 months) or refused treatment with a tyrosine-kinase inhibitor (TKI)
* must have failed (defined as incomplete response or relapse) or refused DLI
* Relapse must have occurred ≥ 60 days after transplant
* Prior DLI is allowed, however not within the 30 days before the 1st dose of ALT-803
* Minimum donor chimerism of 10%
* ≥ 18 years of age
* Karnofsky performance status ≥ 70% (appendix II)
* Adequate organ function within 14 days (30 days for cardiac and pulmonary) of enrollment defined as:

  * Creatinine: ≤ 2.0 mg/dL
  * Hepatic: SGOT/SGPT < 5 x upper limit of institutional normal (ULN)
  * Thyroid Function: Thyroid Stimulating Hormone (TSH) within institutional normal range - patients with thyroid disease are eligible if euthyroid on suppressive or replacement therapy
  * Pulmonary: PFTs > 50% of predicted
  * Cardiac: LVEF by ECHO or MUGA > 40%
* Ability to be off prednisone and other immunosuppressive drugs for at least 30 day before first dose of study drug
* Patient agrees to stay within a reasonable distance (i.e. 30 miles) of the study site for the duration of the study treatment and for a minimum of 48 hours after the last dose and has a dedicated care giver as is standard practice for BMT outpatient care
* Women of child bearing potential and men with partners of child bearing potential must agree to use effective contraception during therapy and for 4 months after completion of therapy
* Voluntary written consent

Exclusion Criteria:

* Post-transplant lymphoproliferative diseases (often referred to as EBV-associated lymphomas)
* Known active CNS leukemia or lymphoma - patients with previously treated CNS disease is permitted if neurologically stable with no ongoing or anticipated need for steroid therapy are eligible
* Ongoing active acute or chronic GVHD requiring immunosuppressive therapy or signs of aGVHD or cGVHD requiring treatment
* Pregnant or lactating - Women of child bearing potential must have a negative pregnancy test within 14 days of study treatment start
* Class II or greater New York Heart Association Functional Classification criteria (appendix II) or serious cardiac arrhythmias likely to increase the risk of cardiac complications of cytokine therapy (e.g. ventricular tachycardia, frequent ventricular ectopy, or supraventricular tachyarrhythmia requiring chronic therapy
* Marked baseline prolongation of QT/QTc interval (e.g. demonstration of a QTc interval greater than 500 milliseconds)
* New progressive pulmonary infiltrates on screening chest x-ray or chest CT scan for which evaluation with bronchoscopy is not feasible. Infiltrates attributed to infection must be stable/improving (with associated clinical improvement) after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections).
* Active bacterial, fungal, or viral infections - all prior infections must have resolved following optimal therapy
* Positive hepatitis C serology or active hepatitis B infection because of the risk of hepatic inflammation and the possible confounding of drug toxicity assessment - chronic asymptomatic viral hepatitis is allowed
* HIV positive because the effect of IL-15 viral loads, HIV immunity, and infectivity of proliferating T cells is unknown
* History of severe asthma, presently on chronic medications (a history of mild asthma not requiring therapy is eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Miller, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (3):
- United States (3):
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Romee R, Cooley S, Berrien-Elliott MM, Westervelt P, Verneris MR, Wagner JE, Weisdorf DJ, Blazar BR, Ustun C, DeFor TE, Vivek S, Peck L, DiPersio JF, Cashen AF, Kyllo R, Musiek A, Schaffer A, Anadkat MJ, Rosman I, Miller D, Egan JO, Jeng EK, Rock A, Wong HC, Fehniger TA, Miller JS. First-in-human phase 1 clinical study of the IL-15 superagonist complex ALT-803 to treat relapse after transplantation. Blood. 2018 Jun 7;131(23):2515-2527. doi: 10.1182/blood-2017-12-823757. Epub 2018 Feb 20. PMID 29463563

RESULTS

PARTICIPANT FLOW:
Groups:
- ALT-803, IV, 1 mcg/kg; ALT-803, IV, 3 mcg/kg; ALT-803, IV, 6 mcg/kg; ALT-803, IV, 10 mcg/kg: Weekly dose of ALT-803 at assigned dose once a week for 4 weeks.
- ALT-803, SQ, 6 mcg/kg: Weekly dose of ALT-803 at assigned dose subcutaneously, once a week for 4 weeks.
- ALT-803, SQ, 10 mcg/kg: Weekly dose of ALT-803 at assigned dose , subcutaneously, once a week for 4 weeks.
Period: Overall Study
Arm/Group | ALT-803, IV, 1 mcg/kg | ALT-803, IV, 3 mcg/kg | ALT-803, IV, 6 mcg/kg | ALT-803, IV, 10 mcg/kg | ALT-803, SQ, 6 mcg/kg | ALT-803, SQ, 10 mcg/kg
Started | 6 | 3 | 4 | 3 | 8 | 9
Completed | 6 | 3 | 4 | 3 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALT-803, IV, 1 mcg/kg | ALT-803, IV, 3 mcg/kg | ALT-803, IV, 6 mcg/kg | ALT-803, IV, 10 mcg/kg | ALT-803, SQ, 6 mcg/kg | ALT-803, SQ, 10 mcg/kg | Total
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 8 | 9 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 1 | 3 | 6 | 6 | 22
  >=65 years | 2 | 1 | 3 | 0 | 2 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 2 | 4 | 5 | 16
  Male | 3 | 2 | 3 | 1 | 4 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 4 | 2 | 7 | 9 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 3 | 4 | 2 | 7 | 9 | 31
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 4 | 3 | 8 | 9 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) Events
Description: The Dose Limiting Toxicity (DLT) is defined as (during first treatment cycle only):
  * any treatment-emergent grade 3 non-hematologic toxicity lasting more than 48 hours (refer to section 6.2.1.1 for full definition)
  * any treatment-emergent grade 4 or 5 non-hematologic toxicity of any duration
  * grade III or IV acute GVHD within 6 weeks after the first ALT-803 dose Maximum Tolerated Dose (MTD) is defined as the dose level where ≤ 1 out of 6 patients has DLT during the first treatment cycle
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ALT-803, IV, 1 mcg/kg | ALT-803, IV, 3 mcg/kg | ALT-803, IV, 6 mcg/kg | ALT-803, IV, 10 mcg/kg | ALT-803, SQ, 6 mcg/kg | ALT-803, SQ, 10 mcg/kg
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 8 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Experiencing Potential Efficacy of ALT 803
Description: The potential efficacy of ALT-803 in this patient population is measured by the responses based on bone marrow examination 1 and 3 months after the last dose of ALT-803.
  Response was defined as follows: for AML and myelodysplastic syndromes (MDS) using the International Working Group modified criteria, non-Hodgkin lymphoma, and multiple myeloma using the International Myeloma Working Group Uniform Response Criteria, and acute lymphoblastic leukemia using protocol-specified criteria.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | ALT-803, IV, 1 mcg/kg | ALT-803, IV, 3 mcg/kg | ALT-803, IV, 6 mcg/kg | ALT-803, IV, 10 mcg/kg | ALT-803, SQ, 6 mcg/kg | ALT-803, SQ, 10 mcg/kg
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 8 | 9
Participants | 0 | 1 | 2 | 0 | 1 | 0

3. Secondary Outcome: Number of Participants With Excessive Toxicity
Description: To evaluate the safety of the ALT-803 when administered on this schedule. Excessive toxicity is defined as having a grade 3-5 non-hematologic, non-relapse and non-infectious toxicity (except fevers alone) based on the NCI's CTCAE version 4.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ALT-803, IV, 1 mcg/kg | ALT-803, IV, 3 mcg/kg | ALT-803, IV, 6 mcg/kg | ALT-803, IV, 10 mcg/kg | ALT-803, SQ, 6 mcg/kg | ALT-803, SQ, 10 mcg/kg
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 8 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Incidence of Acute Graft Versus Host Disease
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | ALT-803, IV, 1 mcg/kg | ALT-803, IV, 3 mcg/kg | ALT-803, IV, 6 mcg/kg | ALT-803, IV, 10 mcg/kg | ALT-803, SQ, 6 mcg/kg | ALT-803, SQ, 10 mcg/kg
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 8 | 9
Participants | 2 | 1 | 1 | 1 | 1 | 3

5. Secondary Outcome: Number of Participants With Incidence of Chronic Graft Versus Host Disease
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | ALT-803, IV, 1 mcg/kg | ALT-803, IV, 3 mcg/kg | ALT-803, IV, 6 mcg/kg | ALT-803, IV, 10 mcg/kg | ALT-803, SQ, 6 mcg/kg | ALT-803, SQ, 10 mcg/kg
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 8 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | ALT-803, IV, 1 mcg/kg | ALT-803, IV, 3 mcg/kg | ALT-803, IV, 6 mcg/kg | ALT-803, IV, 10 mcg/kg | ALT-803, SQ, 6 mcg/kg | ALT-803, SQ, 10 mcg/kg
All-Cause Mortality (participants affected / at risk) | 3/6 | 2/3 | 4/4 | 2/3 | 8/8 | 8/9
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/3 | 0/4 | 0/3 | 6/8 | 6/9
Other Adverse Events (participants affected / at risk) | 4/6 | 2/3 | 2/4 | 2/3 | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALT-803, IV, 1 mcg/kg (N=6) | ALT-803, IV, 3 mcg/kg (N=3) | ALT-803, IV, 6 mcg/kg (N=4) | ALT-803, IV, 10 mcg/kg (N=3) | ALT-803, SQ, 6 mcg/kg (N=8) | ALT-803, SQ, 10 mcg/kg (N=9)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALT-803, IV, 1 mcg/kg (N=6) | ALT-803, IV, 3 mcg/kg (N=3) | ALT-803, IV, 6 mcg/kg (N=4) | ALT-803, IV, 10 mcg/kg (N=3) | ALT-803, SQ, 6 mcg/kg (N=8) | ALT-803, SQ, 10 mcg/kg (N=9)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 2 (2) | 6 (12)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biopsy site oozing (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 3 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dark stools - intermittent (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT01885897/Prot_SAP_000.pdf